CLINICAL TRIAL: NCT06667401
Title: Exploring the Efficacy of Assistive Artificial Intelligence for Ultrasound Guided Regional Anesthesia in Residency Training
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Christopher Fadumiye, MD, Medical College of Wisconsin
Other Study IDs: PRO00052792
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-10

CONDITIONS: Regional Anesthesia
Keywords: Regional anesthesia; Artificial Intelligence; Resident training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- The study will recruit the entire CA1 resident class (n=20): The study will recruit the entire CA1-2 resident class (n=20-30) who have no prior experience with Ultrasound guided regional anesthesia (UGRA) at the Medical College of Wisconsin/Froedtert Hospital. Inclusion criteria include having no prior experience with UGRA. Exclusion criteria include having undergone the regional elective service prior to the inception of the study (CA-2/3 class). No intervention of interest is noted, the cohort will be accessed based on use of the artificial intelligent Ultrasound.
  Interventions: Device: The ScanNav, a novel artificial intelligence device designed to assist in Ultrasound guided regional anesthesia

INTERVENTIONS:
Device: The ScanNav, a novel artificial intelligence device designed to assist in Ultrasound guided regional anesthesia — The ScanNav, a novel artificial intelligence device designed to assist in Ultrasound guided regional anesthesia.We also aim to see of how it enhances teaching and training of residents by experienced regional anesthesia providers. We intend to use surveys/questionnaires of both resident and regional anesthesia provider as they utilize the device in real time.

SUMMARY:
The purpose of this study is to investigate the efficacy of a novel artificial intelligence (AI) device designed to assist in Ultrasound guided regional anesthesia (ScanNav Anatomy Peripheral Nerve Block; ScanNav), in the teaching and training of anesthesiology residents in the subspecialty of regional anesthesia.

DETAILED DESCRIPTION:
Ultrasound-guided regional anesthesia (UGRA) relies on the precise acquisition and interpretation of ultrasound images. The necessary skills to attain this is dependent on the knowledge of the underlying anatomy. Notwithstanding, even experienced anesthesiologists can find this challenging, especially in the setting of anatomical variation, obesity and other potential confounders. This study aims to clarify if The ScanNav, a novel artificial intelligence device designed to assist in UGRA, when utilized with trainees, improves their uptake and training. We also aim to see the relationships of how it enhances teaching and training of residents by experienced regional anesthesia providers.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include any anesthesia resident with no prior experience with UGRA.

Exclusion Criteria:

* Exclusion criteria include any anesthesia resident who has undergone the regional elective service prior to the inception of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The student population includes anesthesia residents in training, and experienced regional anesthesia providers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Qualtric questionaire of participants | From enrollment to the end of device use at 2 weeks.
  Improved teaching and training of anesthesiology residents in the subspecialty of regional anesthesia will be accessed via a questionnaire filled out by participants after use of the device. The questionnaire will access, the type of regional blocks, feasibility of block and ease of teaching with the artificial intelligence Ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data analysed, results, study information and protocol
Supporting Information: Study Protocol, CSR
Time Frame: When published with ICMJE journal and as requested.

REFERENCES:
- [Background] Bowness JS, El-Boghdadly K, Woodworth G, Noble JA, Higham H, Burckett-St Laurent D. Exploring the utility of assistive artificial intelligence for ultrasound scanning in regional anesthesia. Reg Anesth Pain Med. 2022 Jun;47(6):375-379. doi: 10.1136/rapm-2021-103368. Epub 2022 Jan 28. PMID 35091395